CLINICAL TRIAL: NCT05904340
Title: The Efficacy of Social Media Assisted Home-based Transcutaneous Electrical Acupoint Stimulation on Symptoms Associated with Chemotherapy Induced Peripheral Neuropathy in Patients with Breast Cancer
Brief Title: Transcutaneous Electrical Acupoint Stimulation on Symptoms Associated with Chemotherapy Induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 230302
Record Dates: First submitted 2023-05-13; First posted 2023-06-15 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasms; Chemotherapy-induced Peripheral Neuropathy
Keywords: Breast Cancer; Chemotherapy-Induced Peripheral Neuropathy; Transcutaneous Electrical Nerve Stimulation; Transcutaneous Electrical Acupoint Stimulation
MeSH Terms: conditions — Breast Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): The percutaneous nerve discharger (model GM350PP) of APEX low-frequency therapeutic device is used for transcutaneous electrical nerve stimulation of acupoints. The approved number of medical equipment license for this product is: Department of Health Medical Device No. 006696, and the use mode of intervention measures is P5 Disperse -Dense Modulation mode (discharge frequency 2Hz/wave width 260μs/duration 3sec and discharge frequency 100 Hz/wavewidth 140μs/continuation 3sec alternately, maximum discharge volume 80mA), stimulate Neiguan (PC6), Hegu (LI4), Sanyinjiao (SP6) and Taichong (LR3) points, twice a day, 30 minutes each time, for 4 weeks, the intensity is divided into 10-25 mA for hands and 25-40 mA for feet, depending on personal tolerance Adjust flexibly within the interval, and evaluate the severity of neuropathy symptoms of the test every week.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Control Group (No Intervention): 4 weeks of usual care, including prescribe vitamin B6 or B12 and massage therapy. Assessing the severity of neuropathy symptoms every week.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous Electrical Nerve Stimulation (TENS) uses machines to generate electric current, flows through the skin and conducts to the nerves, triggers a chain reaction of nerves through a new stimulus source, and achieves the effect of pain relief. Using different frequencies and intensities will Produce different effects and trigger different physiological mechanisms.
  Other Names: Transcutaneous Electrical Acupoint Stimulation
  Arms: Test Group

SUMMARY:
Breast cancer ranks first in Taiwan's top ten gynecological cancers. Chemotherapy is a standard treatment method for colorectal cancer and breast cancer, but while destroying cancer cells, it also destroys healthy cells, resulting in side effects. Peripheral neuropathy can lead to peripheral nerve damage and decreased activity, which affects the patient's quality of life. Currently, there is no standard and effective method for treating peripheral neuropathy caused by chemotherapy. Therefore, the purpose of this study is to investigate the effect of percutaneous electrical acupoint stimulation on improving peripheral nerve symptoms in breast cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Breast cancer ranks first in Taiwan's top ten gynecological cancers. Chemotherapy is a standard treatment method for colorectal cancer and breast cancer, but while destroying cancer cells, it also destroys healthy cells, resulting in side effects. Peripheral neuropathy can lead to peripheral nerve damage and decreased activity, which affects the patient's quality of life. Currently, there is no standard and effective method for treating peripheral neuropathy caused by chemotherapy. Therefore, the purpose of this study is to investigate the effect of percutaneous electrical acupoint stimulation on improving peripheral nerve symptoms in breast cancer patients undergoing chemotherapy. An experimental study design will be adopted. A convenient sample of 86 patients with breast cancer who completed the chemotherapy course within one month will be recruited from outpatient clinics of a medical center in the middle district of Taiwan. Patients who are eligible and agree to participate will be randomly assigned to the transcutaneous electrical acupoint stimulation group or the control group. The transcutaneous electrical acupoint stimulation group will receive 4 weeks of transcutaneous electrical acupoint stimulation intervention, while the control group will not receive any measures related to this study. Data from both groups will be collected at the time of admission, the 1st week, the 2nd week, the 3rd week, and the 4th week. The study instruments include the cancer treatment-related quality of life neurotoxicity assessment subscale, Total Neuropathy Score clinical version, Brief Pain Inventory interference items scores and hand and foot pain Numerical Rating Scale. The obtained data will be statistically analyzed using SPSS software. The baseline equilibrium of the subjects' demographic and disease characteristics will be examined by the Chi-square test and independent sample T-test. For the main outcome variable Neurotoxicity Subscale and the Numerical Rating Scale for Hand and Foot Pain, generalized estimating equations were used to analyze the effects of between-group, time-to-group, and time-interaction effects. One-way analysis of variance (The Analysis of Variance, ANOVA) to examine intra- and inter-group differences between the clinical version of the Integrated Neuropathy Score and the Simple Pain Scale Interference Item score pretest and posttest (week 4).

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosed with breast cancer for the first time by a physician.
2. Patients who have completed chemotherapy or postoperative adjuvant chemotherapy within 3 months, and the chemotherapy drugs used are paclitaxel, vinblastine or platinum drugs.
3. Patients who have been evaluated by doctors as peripheral neuropathy caused by chemotherapy, and whose symptoms persist after completing chemotherapy.
4. Peripheral sensory or peripheral motor neuropathy grade ≥ 2 in general toxicity criteria (NCI-CTCAE).
5. Those who have clear consciousness and can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. Patients suffering from carcinoma in situ.
2. Patients suffering from stage IV cancer.
3. Patients suffering from metastatic cancer.
4. Patients receiving peripheral neuropathy drugs (Duloxetine)
5. Patients receiving acupoint stimulation therapy.
6. Patients who are allergic to silicone patches.
7. Patients with cardiac pacemakers.
8. Patients suffering from diabetic peripheral neuropathy.
9. Patients suffering from peripheral neuropathy of acquired immunodeficiency syndrome.
10. Patients receiving treatment for mental illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity, FACT/GOG-NTX | pre-intervention.
  sub-scale involve Sensory, motor, auditory and functional impairments, which can reflect the situation that the patient was troubled by symptoms in the past 7 days, a total of 11 items. Record answers in "item response" column. If missing, mark with an X. Perform reversals as indicated, and sum individual items to obtain a score. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered.This produces the subscale score. The higher the score, the better the QOL.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity, FACT/GOG-NTX | up to 4 weeks.
  sub-scale involve Sensory, motor, auditory and functional impairments, which can reflect the situation that the patient was troubled by symptoms in the past 7 days, a total of 11 items. Record answers in "item response" column. If missing, mark with an X. Perform reversals as indicated, and sum individual items to obtain a score. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered.This produces the subscale score. The higher the score, the better the QOL.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity, FACT/GOG-NTX | immediately after the intervention
  sub-scale involve Sensory, motor, auditory and functional impairments, which can reflect the situation that the patient was troubled by symptoms in the past 7 days, a total of 11 items. Record answers in "item response" column. If missing, mark with an X. Perform reversals as indicated, and sum individual items to obtain a score. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered.This produces the subscale score. The higher the score, the better the QOL.

SECONDARY OUTCOMES:
hand and foot pain Numerical Rating Scale | pre-intervention.
  Questions and answers on the severity of symptoms of neuropathic pain in the hands and feet, including burning pain, pins and needles, numbness, loss of sensation, evoked pain, such as touching cold objects, on a numerical scale from 0 to 10, where 0 indicates no symptoms and 1 -3 indicates mild symptoms, 4-6 indicates moderate symptoms, 7-10 indicates severe symptoms, and higher scores indicate more severe symptoms. Please fill in the most uncomfortable parts of your hands and feet, and circle or mark a number on each spectrum to express the answer that applies to you in the past 24 hours.
hand and foot pain Numerical Rating Scale | up to 4 weeks.
  Questions and answers on the severity of symptoms of neuropathic pain in the hands and feet, including burning pain, pins and needles, numbness, loss of sensation, evoked pain, such as touching cold objects, on a numerical scale from 0 to 10, where 0 indicates no symptoms and 1 -3 indicates mild symptoms, 4-6 indicates moderate symptoms, 7-10 indicates severe symptoms, and higher scores indicate more severe symptoms. Please fill in the most uncomfortable parts of your hands and feet, and circle or mark a number on each spectrum to express the answer that applies to you in the past 24 hours.
hand and foot pain Numerical Rating Scale | immediately after the intervention.
  Questions and answers on the severity of symptoms of neuropathic pain in the hands and feet, including burning pain, pins and needles, numbness, loss of sensation, evoked pain, such as touching cold objects, on a numerical scale from 0 to 10, where 0 indicates no symptoms and 1 -3 indicates mild symptoms, 4-6 indicates moderate symptoms, 7-10 indicates severe symptoms, and higher scores indicate more severe symptoms. Please fill in the most uncomfortable parts of your hands and feet, and circle or mark a number on each spectrum to express the answer that applies to you in the past 24 hours.
Total Neuropathy Score clinical version | pre-intervention.
  The test consists of 7 items including motor, sensory, autonomic symptoms, and muscle strength. Each item is scored on a 5-point scale, with each item ranging from 0 to 4 points. The higher the score, the more severe the peripheral neuropathy.
Total Neuropathy Score clinical version | immediately after the intervention.
  The test consists of 7 items including motor, sensory, autonomic symptoms, and muscle strength. Each item is scored on a 5-point scale, with each item ranging from 0 to 4 points. The higher the score, the more severe the peripheral neuropathy.
Brief Pain Inventory interference items scores | pre-intervention.
  The extent to which pain affects general activity, mood, walking ability, work, relationship, sleep, and enjoyment of life There are 7 questions in total, and each question is scored with 11 points. Each question ranges from 0 (not affected) to 10 (completely affected). The higher the score, the more pain affects life. more serious interference.
Brief Pain Inventory interference items scores | immediately after the intervention.
  The extent to which pain affects general activity, mood, walking ability, work, relationship, sleep, and enjoyment of life There are 7 questions in total, and each question is scored with 11 points. Each question ranges from 0 (not affected) to 10 (completely affected). The higher the score, the more pain affects life. more serious interference.

CONTACTS AND LOCATIONS:
Overall Officials: WANG, PHD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess J, Ferdousi M, Gosal D, Boon C, Matsumoto K, Marshall A, Mak T, Marshall A, Frank B, Malik RA, Alam U. Chemotherapy-Induced Peripheral Neuropathy: Epidemiology, Pathomechanisms and Treatment. Oncol Ther. 2021 Dec;9(2):385-450. doi: 10.1007/s40487-021-00168-y. Epub 2021 Oct 16. PMID 34655433
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Cavaletti G, Cornblath DR, Merkies ISJ, Postma TJ, Rossi E, Frigeni B, Alberti P, Bruna J, Velasco R, Argyriou AA, Kalofonos HP, Psimaras D, Ricard D, Pace A, Galie E, Briani C, Dalla Torre C, Faber CG, Lalisang RI, Boogerd W, Brandsma D, Koeppen S, Hense J, Storey D, Kerrigan S, Schenone A, Fabbri S, Valsecchi MG; CI-PeriNomS Group; Mazzeo A, Pace A, Pessino A, Schenone A, Toscano A, Argyriou AA, Brouwer B, Frigeni B, Piras B, Briani C, Dalla Torre C, Dominguez Gonzalez C, Faber CG, Tomasello C, Binda D, Brandsma D, Cortinovis D, Psimaras D, Ricard D, Storey D, Cornblath DR, Galie E, Lindeck Pozza E, Rossi E, Vanhoutte EK, Lanzani F, Pastorelli F, Altavilla G, Cavaletti G, Granata G, Kalofonos HP, Ghignotti I, Merkies ISJ, Bruna J, Hense J, Heimans JJ, Mattavelli L, Padua L, Reni L, Bakkers M, Boogerd M, Campagnolo M, Cazzaniga M, Eurelings M, Leandri M, Lucchetta M, Penas Prado M, Russo M, Valsecchi MG, Piatti ML, Alberti P, Bidoli P, Grant R, Plasmati R, Velasco R, Lalisang RI, Meijer RJ, Fabbri S, Dorsey SG, Galimberti S, Kerrigan S, Koeppen S, Postma TJ, Boogerd W, Grisold W. The chemotherapy-induced peripheral neuropathy outcome measures standardization study: from consensus to the first validity and reliability findings. Ann Oncol. 2013 Feb;24(2):454-462. doi: 10.1093/annonc/mds329. Epub 2012 Aug 21. PMID 22910842
- [Background] Cavaletti G, Jann S, Pace A, Plasmati R, Siciliano G, Briani C, Cocito D, Padua L, Ghiglione E, Manicone M, Giussani G; Italian NETox Group. Multi-center assessment of the Total Neuropathy Score for chemotherapy-induced peripheral neurotoxicity. J Peripher Nerv Syst. 2006 Jun;11(2):135-41. doi: 10.1111/j.1085-9489.2006.00078.x. PMID 16787511
- [Background] Cheng HL, Molassiotis A. Longitudinal validation and comparison of the Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life-Chemotherapy-Induced Peripheral Neuropathy Questionnaire (EORTC QLQ-CIPN20) and the Functional Assessment of Cancer-Gynecologic Oncology Group-Neurotoxicity subscale (FACT/GOG-Ntx). Asia Pac J Clin Oncol. 2019 Feb;15(1):56-62. doi: 10.1111/ajco.13000. Epub 2018 Jun 5. PMID 29873180
- [Background] Ger LP, Ho ST, Sun WZ, Wang MS, Cleeland CS. Validation of the Brief Pain Inventory in a Taiwanese population. J Pain Symptom Manage. 1999 Nov;18(5):316-22. doi: 10.1016/s0885-3924(99)00087-1. PMID 10584454
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hou L, Gu F, Gao G, Zhou C. Transcutaneous electrical acupoint stimulation (TEAS) ameliorates chemotherapy-induced bone marrow suppression in lung cancer patients. J Thorac Dis. 2017 Mar;9(3):809-817. doi: 10.21037/jtd.2017.03.12. PMID 28449490
- [Background] Hou L, Zhou C, Wu Y, Yu Y, Hu Y. Transcutaneous electrical acupoint stimulation (TEAS) relieved cancer-related fatigue in non-small cell lung cancer (NSCLC) patients after chemotherapy. J Thorac Dis. 2017 Jul;9(7):1959-1966. doi: 10.21037/jtd.2017.06.05. PMID 28839994
- [Background] Hung HW, Liu CY, Chen HF, Chang CC, Chen SC. Impact of Chemotherapy-Induced Peripheral Neuropathy on Quality of Life in Patients with Advanced Lung Cancer Receiving Platinum-Based Chemotherapy. Int J Environ Res Public Health. 2021 May 26;18(11):5677. doi: 10.3390/ijerph18115677. PMID 34073174
- [Background] Iravani S, Kazemi Motlagh AH, Emami Razavi SZ, Shahi F, Wang J, Hou L, Sun W, Afshari Fard MR, Aghili M, Karimi M, Rezaeizadeh H, Zhao B. Effectiveness of Acupuncture Treatment on Chemotherapy-Induced Peripheral Neuropathy: A Pilot, Randomized, Assessor-Blinded, Controlled Trial. Pain Res Manag. 2020 Jun 29;2020:2504674. doi: 10.1155/2020/2504674. eCollection 2020. PMID 32676134
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Kerckhove N, Collin A, Conde S, Chaleteix C, Pezet D, Balayssac D. Long-Term Effects, Pathophysiological Mechanisms, and Risk Factors of Chemotherapy-Induced Peripheral Neuropathies: A Comprehensive Literature Review. Front Pharmacol. 2017 Feb 24;8:86. doi: 10.3389/fphar.2017.00086. eCollection 2017. PMID 28286483
- [Background] Kim, S. Y., & Park, J. S. (2021). The Effect of Self-Acupressure on Peripheral Neuropathy, Disturbance in Daily Activity, and Quality of Life in Breast Cancer Patients undergoing Chemotherapy. Asian Oncology Nursing, 21, 129-139. http://www.dbpia.co.kr/journal/articleDetail?nodeId=NODE10606983
- [Background] Oldenmenger WH, de Raaf PJ, de Klerk C, van der Rijt CC. Cut points on 0-10 numeric rating scales for symptoms included in the Edmonton Symptom Assessment Scale in cancer patients: a systematic review. J Pain Symptom Manage. 2013 Jun;45(6):1083-93. doi: 10.1016/j.jpainsymman.2012.06.007. Epub 2012 Sep 25. PMID 23017617
- [Background] Puskulluoglu M, Tomaszewski KA, Grela-Wojewoda A, Pacholczak-Madej R, Ebner F. Effects of Transcutaneous Electrical Nerve Stimulation on Pain and Chemotherapy-Induced Peripheral Neuropathy in Cancer Patients: A Systematic Review. Medicina (Kaunas). 2022 Feb 14;58(2):284. doi: 10.3390/medicina58020284. PMID 35208610
- [Background] Rossoff, J., & Mithal, L. B. (2018). Initial Management of Fever and Neutropenia: A Practical Approach. Clinical Pediatric Emergency Medicine, 19(2), 145-152.
- [Background] Salat K. Chemotherapy-induced peripheral neuropathy-part 2: focus on the prevention of oxaliplatin-induced neurotoxicity. Pharmacol Rep. 2020 Jun;72(3):508-527. doi: 10.1007/s43440-020-00106-1. Epub 2020 Apr 28. PMID 32347537
- [Background] Siregar, E., Herawati, L., Runjati, & Erisna, M. (2020). The Effect ofAcupressure and Acupunture as Natural Induction Methods for Spontaneous Labor: A Systematic Review. International Journal of Nursing and Health Services, 3(6), 743-753. https://doi.org/http://doi.org.10.35654/ijnhs.v3i6.361
- [Background] Song SY, Park JH, Lee JS, Kim JR, Sohn EH, Jung MS, Yoo HS. A Randomized, Placebo-Controlled Trial Evaluating Changes in Peripheral Neuropathy and Quality of Life by Using Low-Frequency Electrostimulation on Breast Cancer Patients Treated With Chemotherapy. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420925519. doi: 10.1177/1534735420925519. PMID 32493088
- [Background] Tsai CH, Lin YH, Li YS, Ho TL, Hoai Thuong LH, Liu YH. Integrated Medicine for Chemotherapy-Induced Peripheral Neuropathy. Int J Mol Sci. 2021 Aug 26;22(17):9257. doi: 10.3390/ijms22179257. PMID 34502166
- [Background] Wong R, Major P, Sagar S. Phase 2 Study of Acupuncture-Like Transcutaneous Nerve Stimulation for Chemotherapy-Induced Peripheral Neuropathy. Integr Cancer Ther. 2016 Jun;15(2):153-64. doi: 10.1177/1534735415627926. Epub 2016 Apr 29. PMID 27130723
- [Background] Xie J, Chen LH, Ning ZY, Zhang CY, Chen H, Chen Z, Meng ZQ, Zhu XY. Effect of transcutaneous electrical acupoint stimulation combined with palonosetron on chemotherapy-induced nausea and vomiting: a single-blind, randomized, controlled trial. Chin J Cancer. 2017 Jan 10;36(1):6. doi: 10.1186/s40880-016-0176-1. PMID 28069044
- [Background] Zajaczkowska R, Kocot-Kepska M, Leppert W, Wrzosek A, Mika J, Wordliczek J. Mechanisms of Chemotherapy-Induced Peripheral Neuropathy. Int J Mol Sci. 2019 Mar 22;20(6):1451. doi: 10.3390/ijms20061451. PMID 30909387